CLINICAL TRIAL: NCT02653989
Title: An International, Phase 2, Open-Label, Efficacy and Safety Study of MDV9300 in Patients With an Incomplete Response Following Salvage Therapy or Autologous Stem Cell Transplantation for Relapsed or Refractory CD20+ Diffuse Large B-Cell Lymphoma
Brief Title: Efficacy and Safety Study of MDV9300 in Patients With Relapsed or Refractory Diffuse Large B-cell Lymphoma (DLBCL)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDV9300-01
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Primary Mediastinal Large B-cell Lymphoma; Transformed Indolent Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDV9300 (Experimental)
  Interventions: Biological: MDV9300

INTERVENTIONS:
Biological: MDV9300 — MDV9300 will be administered at a dose of 200 mg by intravenous (IV) infusion every 2 weeks until treatment discontinuation criteria are met.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of MDV9300 in patients with relapsed or refractory diffuse large B-cell lymphoma (DLBCL) that have achieved either stable disease or a partial remission following definitive salvage therapy.

Two cohorts of patients will be enrolled: a cohort treated with salvage chemotherapy but considered ineligible for autologous stem cell transplant (ASCT), and a cohort of patients who have received ASCT following salvage chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older and willing and able to provide informed consent;
* Histologically confirmed relapsed or refractory CD20+ DLBCL, transformed indolent lymphoma (follicular or other), or primary mediastinal large B-cell lymphoma;
* Received prior treatment with a standard anthracycline and therapeutic anti-CD20 monoclonal antibody-based regimen;
* For transplant-ineligible patients, salvage therapy just prior to MDV9300 treatment must have resulted in a PR or stable disease;
* For post autologous stem cell transplant (ASCT) patients, salvage therapy plus ASCT just prior to MDV9300 treatment must have resulted in a PR or stable disease;
* Adequate bone marrow reserve as defined per protocol;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1. Patients with stable ECOG scores of 2 may be allowed with medical monitor approval.

Exclusion Criteria:

* Burkitt, mantle cell, follicular, or mucosa-associated lymphoid tissue lymphoma
* History of serious autoimmune disease;
* History of central nervous system involvement of lymphoma;
* Prior therapy with agents targeting immune coinhibitory receptors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2018-06 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Best overall response rate | no later than 6 months after the last patient is enrolled in a cohort
  Defined as the proportion of patients in the intent-to-treat population with a complete response (CR) or partial response (PR) attributable to study treatment, as assessed by the independent review committee (IRC).

SECONDARY OUTCOMES:
Duration of response (for responders) | no later than 6 months after the last patient is enrolled in a cohort
  Defined as the time from the first objective evidence of CR or PR as assessed by the IRC to the first objective evidence of disease progression or death due to any cause, whichever occurs first.
Progression-free survival | no later than 6 months after the last patient is enrolled in a cohort
  Defined as the time from the date of first study drug infusion to the first objective evidence of disease progression or death due to any cause, whichever occurs first.
Time to response (for responders) | no later than 6 months after the last patient is enrolled in a cohort
  Defined as the time from the date of first study drug infusion to the first objective evidence of CR or PR as assessed by the IRC.
Overall survival | no later than 6 months after the last patient is enrolled in a cohort
  Defined as the time from the date of first study drug infusion to death due to any cause.
Composite of safety | no later than 6 months after the last patient is enrolled in a cohort
  Safety will be evaluated by incidence and severity of adverse events, including serious adverse events and incidence of permanent treatment discontinuation due to adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Nashville, Tennessee, United States